CLINICAL TRIAL: NCT03488797
Title: Web-based Motor Intervention to Increase Health Related Physical Fitness in Children With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other); Robert-Enke-Stiftung (Unknown); Fördergemeinschaft Deutsche Kinderherzzentren e.V (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: GE TUM FSH DHM I 0118
Record Dates: First submitted 2018-03-12; First posted 2018-04-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Congenital Heart Disease; Health Related Physical Fitness; Motor Skills; Cardiovascular Prevention
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Supervised web- and home-based exercise intervention
  Interventions: Behavioral: Supervised web- and home-based exercise intervention
- No Intervention (No Intervention): Control group - Standard of Care
  * Re-assessment 24 weeks (6 month) after enrolment.
  * Afterwards crossover into experimental group

INTERVENTIONS:
Behavioral: Supervised web- and home-based exercise intervention — * The intervention group gets access to a training platform. Every week, 3 training videos of 20 minutes each will be released on that platform with the aim to perform those during the ongoing week.
  * Each exercise session is arranged in a video session with child friendly instructions and executions for the different exercises. The videos serve as a virtual training partner and exercise will be performed simultaneously while watching the video
  * The overall training volume is 72 session calculated from 3 sessions per week over a duration of 24 weeks (6 month)
  Arms: Experimental

SUMMARY:
Children with congenital heart diseases (CHD) often show reduced health related physical fitness as well as limitations in gross and fine motor skills/development. Intervention programs in childhood are still rare and often focus just on the improvement of cardiac outcomes or exercise capacity. Web-based interventions, as a useful alternative to training manuals or supervised training, are cost effective and allow a customization of training times. Primary purpose of this study is to improve health related physical fitness in children with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Ages 10-18 years old.
* CHD with moderate to complex severity according to the ACC criteria.
* Health-related physical fitness <50th percentile (healthy reference).
* German speaking.
* internet availability and an internet-capable device to use the intervention app
* Informed consent of parent/guardian as well as of the child.

Exclusion Criteria:

* Severe Arrhythmias
* Severe Left Heart Failure
* Chromosomal anomalies and/or genetic syndromes.
* Severe physical and/or sensory impairments (hearing, visual, or psychomotor).
* Elective cardiac intervention within the next 6 months following enrollment.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Improvement of health related physical fitness | at 24 weeks
  The FitnessGram® is a fitness test from the Cooper Institute that assesses health-related physical fitness. It uses evidence-based standards to measure functional health status of the musculoskeletal system divided into the components muscular strength, muscular endurance and flexibility. The FitnessGram® includes tests for the upper body and the abdominal/trunk areas. Mean scores were calculated and compared to an actual reference sample of German children and adolescents.

SECONDARY OUTCOMES:
Compliance with the supervised web- and home-based intervention | at 24 weeks
  Participation rate in training sessions (%)
Central/peripheral blood pressure | at 24 weeks
  mean change in mmHg between intervention and control group
Intima media thickness | at 24 weeks
  mean change in mm between intervention and control group
Pulse-wave-velocity | at 24 weeks
  mean change in m/s between intervention and control group
Change in Health-related Quality of Life (KINDL questionnaire) | at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Hager, MD, Principal Investigator — Department of Paediatric Cardiology and Congenital Heart Defects, German heart center of the state of Bavaria (Munich), Technical University of Munich (TUM)
Locations (1):
- Department of Paediatric Cardiology and Congenital Heart Defects, German Heart Center of the State Bavaria (Munich), Technical University of Munich (TUM), München, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer M, Brudy L, Fuertes-Moure A, Hager A, Oberhoffer-Fritz R, Ewert P, Muller J. E-Health Exercise Intervention for Pediatric Patients with Congenital Heart Disease: A Randomized Controlled Trial. J Pediatr. 2021 Jun;233:163-168. doi: 10.1016/j.jpeds.2021.01.058. Epub 2021 Jan 29. PMID 33516681
- [Derived] Meyer M, Hreinsdottir A, Hacker AL, Brudy L, Oberhoffer R, Ewert P, Muller J. Web-Based Motor Intervention to Increase Health-Related Physical Fitness in Children With Congenital Heart Disease: A Study Protocol. Front Pediatr. 2018 Aug 27;6:224. doi: 10.3389/fped.2018.00224. eCollection 2018. PMID 30211141